CLINICAL TRIAL: NCT06494748
Title: Evaluating the Efficacy of Artificial Intelligence Models in Predicting Intensive Care Unit Admission Needs
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ICU-retro
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Intensive Care Unit
Keywords: artificial intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anesthesiologists Decision: Intensive Care Unit Follow up need is decided by anesthesiologists.
  Interventions: Other: Follow up Decision
- Artificial Intelligence Decision: Intensive Care Unit Follow up need is decided by Artificial Intelligence
  Interventions: Other: Follow up Decision

INTERVENTIONS:
Other: Follow up Decision — 0: No need to follow up in Intensive Care Unit
  1: Need to follow up in Intensive Care Unit

SUMMARY:
This study aims to evaluate the efficacy of two artificial intelligence (AI) models in predicting the need for ICU admissions. By comparing the AI models' predictions with actual clinical decisions, we aim to determine their accuracy and potential utility in clinical decision support.

DETAILED DESCRIPTION:
Intensive care units (ICUs) are critical components of healthcare systems, providing life-saving care to patients with severe and life-threatening conditions. Timely and accurate prediction of ICU admission needs is essential for improving patient outcomes and optimizing hospital resource allocation. Delayed ICU admissions have been consistently associated with higher morbidity and mortality rates. With the advent of artificial intelligence (AI) in healthcare, there is an opportunity to enhance clinical decision-making by leveraging AI models to predict ICU needs accurately. AI models, such as ChatGPT and Gemini, can process vast amounts of complex data to identify patterns that might not be immediately evident to human clinicians, potentially improving the speed and accuracy of ICU admission decisions.

This is an observational retrospective study. Data were collected from electronic health records (EHRs) from a hospital retrospectively.

Data were extracted from EHRs and included:

Demographic data: Age, gender, and basic patient characteristics. Clinical parameters: Medication information, consultation details, ECG findings, imaging results, comorbid conditions (e.g., diabetes mellitus, hypertension, heart failure, COPD, cerebrovascular events), and laboratory values (e.g., hemoglobin, hematocrit, platelet count, PT, INR, procalcitonin, ALT, AST, bilirubin, sodium, potassium, chloride, glucose, creatinine, urea, albumin, thyroid function tests).

Prediction data: AI model predictions and actual ICU admission decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients consulted for anesthesia regarding intensive care needs
* Patients with sufficient data in the hospital's electronic health record system

Exclusion Criteria:

* Patients with insufficient data in the hospital records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 of both genders who are consulted for anesthesia regarding intensive care needs will be included in the study.
Sampling Method: Probability Sample
Enrollment: 8043 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Intensive Care Unit Need | 1 day
  The primary outcome measure of this study is the accuracy of the predictions made by the artificial intelligence (AI) models, ChatGPT and Gemini, regarding the need for ICU admissions. This will be evaluated by comparing the AI model predictions to the actual clinical decisions made regarding ICU admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Specialist, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided